CLINICAL TRIAL: NCT04393415
Title: the Effect of PRP and Cord Blood in Improving the Symptoms of Covid-19
Brief Title: Using PRP and Cord Blood in Treatment of Covid -19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: covid -19
Record Dates: First submitted 2020-05-15; First posted 2020-05-19 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Virus
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patients receiving LGF (Active Comparator)
  Interventions: Combination Product: stem cells
- patients not receiving LGF nor PRP (No Intervention)
- patients receiving Platelet rich plasma (Active Comparator)
  Interventions: Combination Product: stem cells

INTERVENTIONS:
Combination Product: stem cells — giving stem cells to patients with covid - 19
  Arms: patients receiving LGF; patients receiving Platelet rich plasma

SUMMARY:
covid - 19 is a critical viral infection that affects humans

DETAILED DESCRIPTION:
Covid -19 pandemic started was declared in 2020

ELIGIBILITY:
Inclusion Criteria:

* patients with positive covid -19 and has symptoms and isolated in the hospital

Exclusion Criteria:

* patients with negative test for covid -19

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-08-25 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
the number of patients with positive covid 19 who will improve after receiving stem cells | 2 weeks
  patients with positive covid 19 who will improve after receiving stem cells

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Principal Investigator — Algezeera hospitaland National Research Centre ,Egypt
Locations (1):
- Aljazeera( Al Gazeera) hospital, Giza, Egypt